CLINICAL TRIAL: NCT03383744
Title: Using Stable Isotope Techniques to Monitor and Assess the Vitamin A Status of Children Susceptible to Infection
Brief Title: Using Stable Isotopes to Assess the Effectiveness of Vitamin A Supplementation in Cameroon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Food and Nutrition Research, Yaounde (Other Government)
Collaborators: International Atomic Energy Agency (Other Government)
Responsible Party: Principal Investigator, Medoua Nama Gabriel, Head of Centre, Centre for Food and Nutrition Research, Yaounde
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMR_RAF6047
Record Dates: First submitted 2017-12-16; First posted 2017-12-26 (Actual); Last update posted 2017-12-26 (Actual); Status verified 2017-12

CONDITIONS: Vitamin A Deficiency
MeSH Terms: conditions — Vitamin A Deficiency

STUDY DESIGN:
Intervention Model Description: n subjects received the treatment and then randomly divided in two groups for outcome evaluation after one and three months respectively
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin A supplementation 1 (Experimental): Vitamin A status assessed at Baseline and one month after the administration of 200,000 IU of vitamin A
  Interventions: Dietary Supplement: vitamin A supplementation
- Vitamin A supplementation 3 (Experimental): Vitamin A status assessed at Baseline and three months after the administration of 200,000 IU of vitamin A
  Interventions: Dietary Supplement: vitamin A supplementation

INTERVENTIONS:
Dietary Supplement: vitamin A supplementation — Each child received one capsule of 200,000 IU of vitamin A

SUMMARY:
This is a study to evaluate the effects of vitamin A supplementation program on the vitamin A status of preschool children. All children aged 3-5 years who do not have severe illness and are not planning to move from the study area are eligible. Children whose caregivers agree to sign the consent form will be enrolled in their community and submitted to a longitudinal evaluation of vitamin A status before and after vitamin A supplementation campaign.

Vitamin A status will be assessed by measuring serum retinol, retinol binding protein and vitamin A total body pool size using stable isotope dilution methodology.

DETAILED DESCRIPTION:
Five months after the last supplementation (day 0), an oral dose (2 mg retinol equivalents) of label vitamin A ([2H8]-retinyl acetate) in oil will be administered to 80 eligible children together with a low vitamin A high-fat snack. Fasting venous blood samples (about 7 ml) will be collected into evacuated foil-wrapped blood collection tubes specifically designed for the collection of serum (containing no anticoagulant and metal free) on the mornings of days 0 before the administration of the dose and on day 14 for quantitative estimation of initial vitamin A pool size and determination of potential confounding parameters (CRP, AGP, iron, zinc, malaria, carotenoids and retinoids). About six months after the last supplementation (day 30), each child will received the vitamin A supplement. After 30 days and 90 days, two groups of 40 children (Grp1, Grp2) will respectively received a second dose of labeled vitamin A ([2H4]-retinyl acetate); fasting venous blood samples will be obtained before the administration of the dose and 14 days after dosing for quantitative estimation of final vitamin A pool size and determination of potential confounding parameters.

ELIGIBILITY:
Inclusion Criteria:

* Children will be included if they are in the target age range (36-59 months), are not planning to move from the study area for the duration of the study and do not have severe illness at the time of enrolment

Exclusion Criteria:

* Exclusion criteria will generally include the following conditions: severe anaemia, severe acute malnutrition, obesity, or clinically defined severe illness, such as dehydration, severe diarrhoea, malaria or severe respiratory illness

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 104 (Actual)
Dates: Start 2015-10-05 (Actual); Primary Completion 2016-03-23 (Actual); Study Completion 2016-07-29 (Actual)

PRIMARY OUTCOMES:
Change in vitamin A status at one month | One month after vitamin A supplementation
  Change from Baseline vitamin A total body stores at one month
Change in vitamin A status at 3 months | 3 months after vitamin A supplementation
  Change from Baseline vitamin A total body stores at 3 months

REFERENCES:
- [Derived] Imdad A, Mayo-Wilson E, Haykal MR, Regan A, Sidhu J, Smith A, Bhutta ZA. Vitamin A supplementation for preventing morbidity and mortality in children from six months to five years of age. Cochrane Database Syst Rev. 2022 Mar 16;3(3):CD008524. doi: 10.1002/14651858.CD008524.pub4. PMID 35294044